CLINICAL TRIAL: NCT05175157
Title: Assessment of "Gut Feelings" Accuracy Regarding the Effect of Professional Experience in General Practitioners in Clinical Decision Making
Acronym: EGFGP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0359 (EGFGP)
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Gut Feelings

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General practitioner: Answer the Gut Fellings questionnaire
  Interventions: Other: Gut Fellings questionnaire
- Internal: Answer the Gut Fellings questionnaire
  Interventions: Other: Gut Fellings questionnaire

INTERVENTIONS:
Other: Gut Fellings questionnaire — Answer the Gut Fellings questionnaire

SUMMARY:
Knowledge, experience and professional development limit the risk of diagnostic error for the clinician in daily practice. However, research has shown that other non-analytical factors are involved in clinical decision making. Intuition (or "gut feelings") is a subjective element involved in medical decision-making, and its place and relevance are being explored. The concept of "gut feelings" comes from General Practitioners (GPs) themselves and their description of their own practice. Several studies have shown its place in medical decision-making models, particularly in the face of diagnostic uncertainty.

A questionnaire used as a standardized measurement tool for gut feelings was created to address this issue. The Gut Feelings Questionnaire (GFQ) has been translated into French, German and Polish during a standardized linguistic validation procedure. It is currently validated and available in five languages. The QGF has been tested and validated in clinical practice by Belgian, French and Dutch physicians. Its feasibility has been evaluated in these three health systems.

The Gut Feelings Questionnaire was used in a prospective study to determine the accuracy of the sense of alarm in patients consulting their GP for chest pain and/or dyspnea. But the role of the practitioner's experience has not been studied: is the gut feeling more accurate in experienced GPs than in first semester interns in general practice?

ELIGIBILITY:
Inclusion Criteria:

- GP population: General practitioners established for more than 3 years

- Intern population: Interns in general medicine in the first year of the third cycle of the diploma of specialized studies in general medicine

Exclusion Criteria:

- For the 2 populations: Refusal to participate

- Intern population: Interns in the second and third year of the diploma of specialized studies in general medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * General practitioners established for more than 3 years
  * Interns in the first year of the third cycle of the diploma of specialized studies in general medicine of the Universities of Brest and Rouen
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Error assessment | Day 1
  Gut Feelings Questionnaire response score comparaison for each of 12 clinical vignettes. Gut Feelings Questionnaire is a 10-item questionnaire based on the definitions of the sense of alarm and the sense of reassurance. The purpose of the Gut Feelings Questionnaire is to determine the presence or absence of gut feelings in the diagnostic reasoning. These gut feelings are defined as a 'sense of alarm' and a 'sense of reassurance'. A 'sense of alarm' implies that a GP worries about a patient's health status, even though he/she has found no specific indications yet; it is a sense that 'there's something wrong here'. A 'sense of reassurance' means that a GP feels secure about the further management and course of a patient's problem, even though he/she may not be certain about the diagnosis: everything fits in.

SECONDARY OUTCOMES:
Types of professional activity of installed GPs | Day 1
  To study the relationship between professional variables and GFQ response score errors in the GP population. Professional variables are be : University training supervisor (yes/no); type of activity (group of physicians, alone, multiprofessional group); place of practice (town of <2000 inhabitants, between 2000 and 5000, over 5000); number of years of practice in general medicine.
Type of care | Day 1
  Care proposed at the end of each clinical vignette (answers to question n°11 of the questionnaire)
Practitioner's orientation | Day 1
  Items highlighted by each participant within the clinical vignette that contributed to the practitioner's orientation (identification of a sense of alarm or a sense of reassurance) to complete the Gut Fellings Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Marie BARAIS, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After result publication
Access Criteria: The data that will support the findings of this study will be available when the findings will be published in a perreview journal, from the corresponding author, upon reasonable request